CLINICAL TRIAL: NCT06894069
Title: Effect of Intentional Extrusion of an Intracanal Corticosteroid Solution on Post Endodontic Treatment Pain: a Randomized Clinical Trial
Brief Title: Intracanal Dexamethasone Extrusion and Postoperative Endodontic Pain
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Renad Hazem Khanfer, Doctor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10/2023/ 32001
Record Dates: First submitted 2025-01-23; First posted 2025-03-25 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Post Operative Pain Control; Endodontic Treatment
Keywords: Root canal treatment; Post-operative pain; Corticosteroids; Dexamethasone; Randomised controlled trial
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DXM (Experimental): Patients in this group will receive a standard root canal treatment but with the extra step of extruding a Dexamethasone (DXM) solution through the root canals to the periradicular tissues prior to obturation.
  Interventions: Drug: Dexamethasone
- Saline (Placebo Comparator): Patients in this group will receive a standard root canal treatment with saline used as the final irrigating solution prior to obturation.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone — a 2 ml solution of dexamethasone (3.3mg/ml) will be flushed in the root canal and intentionally extruded to the periradicular tissues to assess its potnetial sedative effect
  Arms: DXM
Other: Placebo — 2ml of normal saline will be used as placebo to be flushed and extruded through the canals to the periradicular tissues
  Arms: Saline

SUMMARY:
The aim of this research is to assess the effect of intentionally extruding a corticosteroid intracanal solution into the periapical tissues on the postoperative pain after root canal treatment in patients with symptomatic irreversible pulpitis and symptomatic apical periodontitis (SIP/SAP). The main question it aims to answer: Is there an analgesic effect of extruding an intracanal solution of DXA into the periapical tissues in patients diagnosed with SIP/SAP? Researchers will compare dexamethasone to a placebo to see if the extrusion dexamethasone works in reducing post-endodontic treatment pain.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of irreversible pulpits with symptomatic apical periodontitis
* Adult patients (aged 18 - 70)
* Healthy patients or those with a well-controlled disease (ASA I & II)

Exclusion Criteria:

* A diagnosis of necrotic pulp, or normal apical tissues
* Patients with a severe systemic disease (ASA III or higher)
* Patients who received analgesics12 hours before presentation
* Previously treated/initiated Endodontics treatment on the same tooth
* Unopposed teeth
* Third molar teeth
* Non-restorable teeth
* Periodontally compromised teeth
* Pregnant or lactating patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain following root canal treatment | at 12, 24, 48 and 72 hours after completing the treatment
  The outcome measure is patient-reported pain following root canal treatment. Patients will be given a questionnaire to complete, on 4 different time intervals following the completion of their root canal treatment (12, 24, 48 and 72 h). For each time interval, patients will be asked to fill out:
  1. their perceived pain level on a standard 100mm visual-analogue scale, with pain values ranging from zero (no pain at all) and ascending gradually until 100 (worst imagined pain).
  2. Whether they needed to take any analgesics. In this case, details about the type, route, dose and timing of the analgesic taken will have to be filled out

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol